CLINICAL TRIAL: NCT05987566
Title: Chronobiology of Meal Timing: Effects on Vascular and Renal Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: HM20026660
Record Dates: First submitted 2023-07-31; First posted 2023-08-14 (Actual); Last update posted 2024-03-19 (Actual); Status verified 2024-03

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Morning Meal Challenge (Experimental)
  Interventions: Other: Morning meal challenge
- Late Night Meal Challenge (Experimental)
  Interventions: Other: Evening meal challenge

INTERVENTIONS:
Other: Morning meal challenge — A Western-style diet meal which will be individualized for caloric consumption by estimated total daily energy expenditure eaten after 1 hour of waking up in the morning
  Arms: Morning Meal Challenge
Other: Evening meal challenge — A Western-style diet meal which will be individualized for caloric consumption by estimated total daily energy expenditure eaten within 1 hour of going to bed
  Arms: Late Night Meal Challenge

SUMMARY:
The purpose of this study us to investigate the effects of mistimed eating on blood pressure, kidney function and vascular function.

DETAILED DESCRIPTION:
Despite advancements in pharmacologic antihypertensives, hypertension currently affects 1 in 3 Americans and accounts for more than $50 billion of health care spending. Importantly, hypertension is the leading cause of cardiovascular (CVD) and kidney diseases (CKD). As a result, the AHA/ACC lowered the diagnostic criteria for hypertension to encourage earlier preventative lifestyle intervention. There is a critical need to identify and implement novel lifestyle interventions in individuals with early-stage hypertension to prevent the subsequent development of CVD and CKD. Chronotherapy that aligns behavioral cues (such as time of eating) with the body's internal biological clocks, has gained much attention as a potential strategy to prevent and manage hypertension, however, the underlying mechanisms are not yet fully understood. The purpose of this study is to investigate the effects of mistimed eating on blood pressure, kidney function and vascular function.

ELIGIBILITY:
Inclusion Criteria:

* Men and Women aged 18-45 years
* Elevated (SBP 120-129; DBP <80 mmHg) or stage 1 hypertension (SBP 130-139; DBP 80-89 mmHg)

Exclusion Criteria:

* History of chronic disease (CV, lung, cancer, renal, sleep apnea, diabetes, autoimmune)
* Anti-hypertensive medication use
* Currently pregnant or lactating
* Current shift worker
* Travel >3 time zones four weeks before the start of the study or during the study
* Insomnia
* Practiced intermittent fasting in past six months
* Current nicotine use
* Current hormone replacement therapy
* Current melatonin use
* Current use of antioxidants and unwilling to stop taking them for the duration of the study
* Unable to provide informed consent

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2023-09-11 (Actual); Primary Completion 2024-03-06 (Actual); Study Completion 2024-03-06 (Actual)

PRIMARY OUTCOMES:
Urinary sodium excretion and markers of kidney injury | 24 hours
  Day and nocturnal urinary sodium, NGAL and KIM-1

SECONDARY OUTCOMES:
24hr ambulatory blood pressure | 24 Hours
  Day and nocturnal ambulatory blood pressure
Macrovascular function | At baseline and after each 24hour experimental arm
  Brachial artery endothelial function assessed by flow mediated dilation
Microvascular function | At baseline and after each 24hour experimental arm
  Skin blood flow response to local heating measured by laser doppler flowmetry

CONTACTS AND LOCATIONS:
Overall Officials: Danielle Kirkman, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth Univesity, Richmond, Virginia, United States

IPD SHARING:
Plan to Share IPD: No